CLINICAL TRIAL: NCT02093364
Title: A Focused Registry to Document the Use of the Short- or Long-stemmed Radial Head Prosthesis (RHP)
Status: Withdrawn | Type: Observational
Why Stopped: No participants enrolled
Sponsor: AO Clinical Investigation and Publishing Documentation (Other)
Responsible Party: Sponsor
Organization: AO Innovation Translation Center (Other)
Other Study IDs: FR Radial Head Prosthesis
Record Dates: First submitted 2014-03-18; First posted 2014-03-21 (Estimated); Last update posted 2020-08-12 (Actual); Status verified 2020-08

CONDITIONS: Fracture of the Radial Head Which is Not Amendable to an Adequate Osteosynthesis; Post-traumatic Deformity or Arthroses; Failed Open Reduction Internal Fixation (ORIF) of a Radial Head Fracture; Failed Conservative Radial Head Fracture Treatment
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this focused registry is to evaluate the clinical implications of the RHP position (relative to the articulations) regarding functional and radiographic parameters in patients treated with the RHP with a straight and curved stem.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Use of a short-or long-stemmed DePuy Synthes Radial Head Prosthesis due to any of the following indications:

  * Fresh fracture of the radial head which is not amendable to an adequate -steosynthesis
  * Post-traumatic deformity or arthroses
  * Failed open reduction internal fixation (ORIF)
  * Failed conservative radial head fracture treatment
* Informed consent obtained, i.e.:

  * Ability to understand the content of the patient information / Informed Consent Form
  * Willingness and ability to participate in the clinical investigation according to the Clinical Investigation Plan (CIP)
  * Signed and dated Ethics Committee (EC) / Institutional Review Board (IRB) approved written informed consent

Exclusion Criteria:

* Active infection at the affected elbow
* Any not medically managed severe systemic disease
* Pregnancy
* Prisoner
* Recent history of substance abuse (ie, recreational drugs, alcohol) that would preclude reliable assessment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care centers
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2015-07; Primary Completion 2015-12 (Estimated); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Evaluation of the functional outcome | 12 Months
  Elaborate if there is an association between the implant head and stem position (relative to the elbow articulations), functional outcomes and radiological parameters (radiolucency and arthritis) after 1 year in patients treated with a RHP

SECONDARY OUTCOMES:
Evaluation of functional outcome | 24 months
  Elaborate if there is an association between the implant head and stem position (relative to the elbow articulations), functional outcomes and radiological parameters (radiolucency and arthritis) after 2 years
Range of motion | 12 months
  To investigate range of motion of the injured limb as compared to the contralateral side
Adverse events | 12 months
  To evaluate if the related adverse events have an effect on quality of life (EQ5D)